CLINICAL TRIAL: NCT01975337
Title: An Open-label Study to Evaluate the Pharmacokinetics and Safety of a Single Oral Dose of Alisporivir (DEB025) in Subjects With End Stage Renal Disease on Hemodialysis Compared to Matched Healthy Subjects
Brief Title: Pharmacokinetics and Safety of Alisporivir in Subjects With End Stage Renal Disease on Hemodialysis Compared to Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Debiopharm International SA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: CDEB025A2112
Record Dates: First submitted 2013-10-07; First posted 2013-11-04 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Kidney Failure, Chronic
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — alisporivir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- End stage renal disease participants (Experimental): End stage renal disease (ESRD) participants received a single 400 mg (2 x 200 mg capsules) oral dose of alisporivir with food at any time during the 2 hours after completion of hemodialysis on Day 1.
  Interventions: Drug: Alisporivir
- Matched healthy participants (Active Comparator): Healthy participants (matched to those with end stage renal disease by sex, age, weight, and smoking status), received a single 400 mg (2 x 200 mg capsules) oral dose of alisporivir with food on Day 1.
  Interventions: Drug: Alisporivir

INTERVENTIONS:
Drug: Alisporivir — Alisporivir supplied as 200 mg oral capsules in blister packs (7 units per blister pack)
  Other Names: DEB025

SUMMARY:
The primary objective of the study was to compare the single dose pharmacokinetics of alisporivir in subjects with end stage renal disease (ESRD) on hemodialysis to those of matched healthy subjects. The secondary objective was to evaluate the safety and tolerability of a single dose of alisporivir when administered to subjects with ESRD.

ELIGIBILITY:
Inclusion Criteria:

* Provides written informed consent before any assessment is performed
* Matched healthy participants are in good health as determined by past medical history, physical examination, vital signs, laboratory tests, and other assessments
* ESRD participants are on a protocol-defined stable hemodialysis regimen and have no evidence of hepatic decompensation, with vital signs and other tests within protocol-specified limits
* Weighs at least 50 kg
* Is able to communicate well with the investigator, to understand and comply with the requirements of the study.

Exclusion Criteria:

* Has history or current use of over-the-counter medications, dietary supplements, or drugs (including nicotine and alcohol) outside protocol-specified parameters
* Has signs, symptoms or history of any condition that, per protocol or in the opinion of the investigator, might compromise:

  1. the safety or well-being of the participant or study staff;
  2. the safety or well-being of the participant's offspring (such as through pregnancy or breast-feeding);
  3. the analysis of results

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-08; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Observed maximum plasma concentration of alisporivir following drug administration [mass / volume] (Cmax) | Pre-dose (0 hours) and 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 60, and 65 hours post-dose
Area under the plasma concentration-time curve for alisporivir from time zero to time 'infinity' [mass x time / volume] (AUCinf) | Pre-dose (0 hours) and 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 60, and 65 hours post-dose
Area under the plasma concentration-time curve for alisporivir from time zero to the time of the last quantifiable concentration [mass x time / volume] (AUClast) | Pre-dose (0 hours) and 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 60, and 65 hours post-dose

SECONDARY OUTCOMES:
Time to reach peak or maximum concentration of alisporivir following drug administration [time] (Tmax) | Pre-dose (0 hours) and 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 60, and 65 hours post-dose
The terminal elimination half-life [time] (T1/2) for alisporivir | Pre-dose (0 hours) and 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 60, and 65 hours post-dose
Apparent systemic (or total body) clearance from plasma following extravascular administration of alisporivir [volume / time] (CL/F) | Pre-dose (0 hours) and 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 60, and 65 hours post-dose
The apparent volume of distribution during the terminal elimination phase following extravascular administration of alisporivir [volume] (Vz/F) | Pre-dose (0 hours) and 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 60, and 65 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Orlando, Florida, United States